CLINICAL TRIAL: NCT05264480
Title: A Novel Periodontally Accelerated Osteogenic Orthodontics (PAOO) in the Prevention of Buccal Bone Dehiscence in Patients Receiving Orthodontic Therapy- a Randomized Controlled Clinical Trial
Brief Title: The Introduction of a Novel PAOO Technique
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Collaborators: NSK Europe GmbH (Industry)
Responsible Party: Principal Investigator, Pal Nagy, Senior Lecturer, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PIEZO-ORTHO
Record Dates: First submitted 2022-02-20; First posted 2022-03-03 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Bone Loss; Tooth Movement
Keywords: periodontally accelerated osteogenic orthodontics; orthodontic tooth movement; corticotomy; bone augmentation
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Intervention Model Description: Subjects are randomly allocated either to test (bone augmentation with corticotomy) or control (without corticotomy) groups
Who Masked: Outcomes Assessor
Masking Description: The persons responsible to measure on the cephalogramms and CBCTs are blinded to the study design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Test patients receive bone augmentation and selective decorticalisation (corticotomy) and 1 week postop. OTM.
  Interventions: Procedure: Bone augmentation with minimally invasive corticotomy (piezotomy)
- Control group (Active Comparator): Control subjects receive bone augmentation without decorticalisation (corticotomy) and 1 week postop. OTM.
  Interventions: Procedure: Bone augmentation without corticotomy

INTERVENTIONS:
Procedure: Bone augmentation with minimally invasive corticotomy (piezotomy) — Double layer tunnel flap preparation. Subperiosteally "sticky bone" containing platelet rich fibrin (PRF) and xenograft is utilized for bone augmentation, while supraperiosteally PRF membranes are used for soft tissue augmentation. Trough the vertical releasing incisions a piezosurgical device is used to perform corticotomy. 1 week after surgery OTM is initiated.
  Arms: Test group
Procedure: Bone augmentation without corticotomy — Double layer tunnel flap preparation. Subperiosteally "sticky bone" containing platelet rich fibrin (PRF) and xenograft is utilized for bone augmentation, while supraperiosteally PRF membranes are used for soft tissue augmentation. Corticotomy is not performed in this group. 1 week after surgery OTM is initiated.
  Arms: Control group

SUMMARY:
The aim of this study is to evaluate in a prospective, randomized, controlled clinical trail the effectiveness of preorthodontic piezotomy combined with a buccal bone augmentation (in other name periodontlly accelerated osteogenic orthodontics: PAOO)in the prevention of gingival recession, and in the acceleration of orthodontic tooth movement (OTM).

DETAILED DESCRIPTION:
Patients presenting teeth crowding in mandibulary or maxillary front area, without ongoing periodontal disease, who require OTM with incisor proclination, are included in the study. Patients are randomly allocated into test and control groups. Individuals in both groups receive before OTM a buccal bone augmentation in order to further increase the bony envelope where to teeth are intended to move. Test subjects receive a selected decorticalistation of the buccal bone with a piezosurgical device (piezotomy), while control patients are augmented without piezotomy. 1 week postsurgical multibond orthodontic appliances are bonded to initiate OTM. Teeth movement are measured on cephalometric X-ray images, where an initial and a final (at the end of the nivellation phase) cephalogramm is compared with each other. Buccal bone dimensions are measured on initial and 6th month's postoperatively CBCT images. The investigators' hypothesis is that the buccal bone thickness can be significantly increased, which might prevent the development of gingival recessions. This means, that in both groups the initial and final bone volumes will be comparable without significant difference. It is also hypothesized that the bone changes will not differ significantly between the two groups. However, piezotomy in the test group might have an additional benefit throughout regional acceleratory phenomenon, reducing the duration of OTM.

ELIGIBILITY:
Inclusion Criteria:

* tooth crowding exceeding a 5mm lack of space (originating from the discrepancy between the overall mesiodostal length of the teeth and the length of the dental arch present at the time of the evaluation)
* thin bone morphotype (buccal width of the cortical layer must be under 1mm)
* incisor proclination in order to eliminate crowding without compensatory extractions.
* informed consent

Exclusion Criteria:

* ongoing periodontitis
* Pregnant women.
* Participation in another clinical study within 30 days prior to study start.
* Alcoholism, drug dependency, heavy smoking (>5 cigarettes/day).
* Known infection with HIV, HBV, or HCV.
* Patients requiring chemo- or radiotherapy.
* Previous or current radiotherapy of the head.
* Uncontrolled or insulin-dependent diabetes mellitus
* Clinically relevant osteoporosis or systemic disease affecting bone metabolism
* Clinically relevant cardiovascular disease e.g., decompensated cardiac insufficiency, hemodynamically relevant heart valve defects, or myocardial infarction during the last three months.
* Clinically relevant blood coagulation disorder.
* Previous or current treatment with systemic corticosteroids (within 2 months prior to screening visit) of more than 5 mg/day prednisone equivalent.
* Previous or current therapy with bisphosphonates at least for 30 days within the last 12 months before screening visit

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Speed of OTM | From the date of orthodontic appliance bonding until the date of documented finalization of nivellation phase of OTM registered by the orthodontic specialist (in weeks), assessed up to maximum of 25 weeks.
  The angle and distance of the movement of the middle incisor are measure on cephalogramms. The values are divided by the elapsed time frame in order to calculate the speed of OTM.

SECONDARY OUTCOMES:
Vertical bone level | 6 months postoperatively
  The distance between the cement-enamel junction and the crestal bone on the buccal aspect of the mandibular anterior teeth.
Horizontal bone levels | 6 months postoperatively
  The buccal bone thickness measured at 4,7 and 9mm distances from the cement-enamel junction of the mandibular anterior teeth. The thickness is measured on CBCT coronal slices.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Windisch, Professor, Study Director — Semmelweis University
Locations (1):
- Semmelweis University Department of Periodontology, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahn HW, Seo DH, Kim SH, Park YG, Chung KR, Nelson G. Morphologic evaluation of dentoalveolar structures of mandibular anterior teeth during augmented corticotomy-assisted decompensation. Am J Orthod Dentofacial Orthop. 2016 Oct;150(4):659-669. doi: 10.1016/j.ajodo.2016.03.027. PMID 27692424
- [Background] Artun J, Krogstad O. Periodontal status of mandibular incisors following excessive proclination. A study in adults with surgically treated mandibular prognathism. Am J Orthod Dentofacial Orthop. 1987 Mar;91(3):225-32. doi: 10.1016/0889-5406(87)90450-1. PMID 3469907
- [Background] Coscia G, Coscia V, Peluso V, Addabbo F. Augmented corticotomy combined with accelerated orthodontic forces in class III orthognathic patients: morphologic aspects of the mandibular anterior ridge with cone-beam computed tomography. J Oral Maxillofac Surg. 2013 Oct;71(10):1760.e1-9. doi: 10.1016/j.joms.2013.04.022. Epub 2013 Jun 15. PMID 23773424
- [Background] Lee KB, Lee DY, Ahn HW, Kim SH, Kim EC, Roitman I. Tooth movement out of the bony wall using augmented corticotomy with nonautogenous graft materials for bone regeneration. Biomed Res Int. 2014;2014:347508. doi: 10.1155/2014/347508. Epub 2014 Aug 27. PMID 25247172
- [Background] Lund H, Grondahl K, Grondahl HG. Cone beam computed tomography evaluations of marginal alveolar bone before and after orthodontic treatment combined with premolar extractions. Eur J Oral Sci. 2012 Jun;120(3):201-11. doi: 10.1111/j.1600-0722.2012.00964.x. PMID 22607336
- [Background] Murphy KG, Wilcko MT, Wilcko WM, Ferguson DJ. Periodontal accelerated osteogenic orthodontics: a description of the surgical technique. J Oral Maxillofac Surg. 2009 Oct;67(10):2160-6. doi: 10.1016/j.joms.2009.04.124. No abstract available. PMID 19761909